CLINICAL TRIAL: NCT05466435
Title: Efficacy of Heavy Slow Resistance Training in Adults With Frozen Shoulder- a Double Blind Randomised Controlled Trial
Brief Title: Heavy Slow Resistance Training in Adults With Frozen Shoulder
Acronym: HSRFSRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, N.A.RAFI AHMED, Principal Investigator, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121
Record Dates: First submitted 2022-07-04; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; Heavy slow resistance; Isometrics; Eccentric exercise; Muscle guarding
MeSH Terms: conditions — Bursitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy Slow Resistance group (Experimental): Heavy slow resistance exercise will be given along with traditional physical therapy program
  Interventions: Other: Heavy Slow Resistance; Other: Control group
- Control group (Placebo Comparator): Traditional physical therapy program will be given to the control group
  Interventions: Other: Control group

INTERVENTIONS:
Other: Heavy Slow Resistance — Heavy slow resistance exercise will be given twice a week for 12 weeks along with traditional physical therapy program
  Arms: Heavy Slow Resistance group
Other: Control group — Traditional physical therapy program only will be given twice a week for 12 weeks

SUMMARY:
The aim of the study is to evaluate the efficacy of Heavy Slow Resistance exercise in patients diagnosed with frozen shoulder using randomized controlled trial design

ELIGIBILITY:
Inclusion Criteria:

* Unilateral painful, restricted active and passive range of motion of the shoulder, with loss of passive external rotation of at least 50% compared to opposite side at 0 deg of abduction
* Symptoms present for at least 3 months
* Normal x-rays on anteroposterior, axillary and lateral views

Exclusion Criteria:

* Severe degeneration, or trauma involving the shoulder
* Inflammatory joint disease affecting the shoulder.
* Pain or disorders of the cervical spine, elbow, wrist, or hand
* Stroke or peripheral nerve neuropathy Injection with corticosteroids in the affected shoulder in the preceding 4 weeks.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Range of motion measurement for external rotation and abduction using clinometer application at week 12 | week 12 from baseline measurement
  The smart phone clinometer is a validated tool to measure range of motion

SECONDARY OUTCOMES:
Quick DASH(Quick Disabilities of the of Arm Shoulder and Hand) | week 12 from baseline measurement
  Quick DASH is an 11 item questionnaire to measure physical function and symptoms in people presenting with one or more disabilities of the arm, shoulder, and hand. The higher the score from 0 to 100 scale the higher the disability.
12-Item Short Form Health Survey (SF-12) | week 12 from baseline measurement
  SF-12 is a 12 item ,self-reported outcome measure for assessing quality of life.
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
The Oxford Shoulder Score(OSS) | week 12 from baseline measurement
  The Oxford Shoulder Score is validated tool for measuring pain and disability caused by shoulder pathology. It has 12 items with a score ranging from 0 to 48 with 48 being the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Ahmed, MPT, Principal Investigator — Ministry of Health, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five years after completing the study

REFERENCES:
- [Background] Jurgel J, Rannama L, Gapeyeva H, Ereline J, Kolts I, Paasuke M. Shoulder function in patients with frozen shoulder before and after 4-week rehabilitation. Medicina (Kaunas). 2005;41(1):30-8. PMID 15687748
- [Background] Mao CY, Jaw WC, Cheng HC. Frozen shoulder: correlation between the response to physical therapy and follow-up shoulder arthrography. Arch Phys Med Rehabil. 1997 Aug;78(8):857-9. doi: 10.1016/s0003-9993(97)90200-8. PMID 9344306
- [Background] Bulgen DY, Binder AI, Hazleman BL, Dutton J, Roberts S. Frozen shoulder: prospective clinical study with an evaluation of three treatment regimens. Ann Rheum Dis. 1984 Jun;43(3):353-60. doi: 10.1136/ard.43.3.353. PMID 6742895
- [Background] Mezian K, Coffey R, Chang KV. Frozen Shoulder(Archived). 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482162/ PMID 29489251
- [Background] Neviaser JS. Adhesive capsulitis and the stiff and painful shoulder. Orthop Clin North Am. 1980 Apr;11(2):327-31. PMID 7001312
- [Background] Chan HBY, Pua PY, How CH. Physical therapy in the management of frozen shoulder. Singapore Med J. 2017 Dec;58(12):685-689. doi: 10.11622/smedj.2017107. PMID 29242941
- [Background] Page MJ, Green S, Kramer S, Johnston RV, McBain B, Chau M, Buchbinder R. Manual therapy and exercise for adhesive capsulitis (frozen shoulder). Cochrane Database Syst Rev. 2014 Aug 26;2014(8):CD011275. doi: 10.1002/14651858.CD011275. PMID 25157702
- [Background] Johnson AJ, Godges JJ, Zimmerman GJ, Ounanian LL. The effect of anterior versus posterior glide joint mobilization on external rotation range of motion in patients with shoulder adhesive capsulitis. J Orthop Sports Phys Ther. 2007 Mar;37(3):88-99. doi: 10.2519/jospt.2007.2307. PMID 17416123
- [Background] Diercks RL, Stevens M. Gentle thawing of the frozen shoulder: a prospective study of supervised neglect versus intensive physical therapy in seventy-seven patients with frozen shoulder syndrome followed up for two years. J Shoulder Elbow Surg. 2004 Sep-Oct;13(5):499-502. doi: 10.1016/j.jse.2004.03.002. PMID 15383804
- [Background] Yoon SH, Lee HY, Lee HJ, Kwack KS. Optimal dose of intra-articular corticosteroids for adhesive capsulitis: a randomized, triple-blind, placebo-controlled trial. Am J Sports Med. 2013 May;41(5):1133-9. doi: 10.1177/0363546513480475. Epub 2013 Mar 18. PMID 23507791
- [Background] Celik D, Kaya Mutlu E. Does adding mobilization to stretching improve outcomes for people with frozen shoulder? A randomized controlled clinical trial. Clin Rehabil. 2016 Aug;30(8):786-94. doi: 10.1177/0269215515597294. Epub 2015 Jul 30. PMID 26229109
- [Background] Maund E, Craig D, Suekarran S, Neilson A, Wright K, Brealey S, Dennis L, Goodchild L, Hanchard N, Rangan A, Richardson G, Robertson J, McDaid C. Management of frozen shoulder: a systematic review and cost-effectiveness analysis. Health Technol Assess. 2012;16(11):1-264. doi: 10.3310/hta16110. PMID 22405512
- [Background] Rangan A, Brealey SD, Keding A, Corbacho B, Northgraves M, Kottam L, Goodchild L, Srikesavan C, Rex S, Charalambous CP, Hanchard N, Armstrong A, Brooksbank A, Carr A, Cooper C, Dias JJ, Donnelly I, Hewitt C, Lamb SE, McDaid C, Richardson G, Rodgers S, Sharp E, Spencer S, Torgerson D, Toye F; UK FROST Study Group. Management of adults with primary frozen shoulder in secondary care (UK FROST): a multicentre, pragmatic, three-arm, superiority randomised clinical trial. Lancet. 2020 Oct 3;396(10256):977-989. doi: 10.1016/S0140-6736(20)31965-6. PMID 33010843
- [Background] Pruimboom L, van Dam AC. Chronic pain: a non-use disease. Med Hypotheses. 2007;68(3):506-11. doi: 10.1016/j.mehy.2006.08.036. Epub 2006 Oct 30. PMID 17071012
- [Background] Donatelli R, Ruivo RM, Thurner M, Ibrahim MI. New concepts in restoring shoulder elevation in a stiff and painful shoulder patient. Phys Ther Sport. 2014 Feb;15(1):3-14. doi: 10.1016/j.ptsp.2013.11.001. Epub 2013 Nov 16. PMID 24315683
- [Background] Maenhout AG, Mahieu NN, De Muynck M, De Wilde LF, Cools AM. Does adding heavy load eccentric training to rehabilitation of patients with unilateral subacromial impingement result in better outcome? A randomized, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1158-67. doi: 10.1007/s00167-012-2012-8. Epub 2012 May 12. PMID 22581193
- [Background] Dejaco B, Habets B, van Loon C, van Grinsven S, van Cingel R. Eccentric versus conventional exercise therapy in patients with rotator cuff tendinopathy: a randomized, single blinded, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2017 Jul;25(7):2051-2059. doi: 10.1007/s00167-016-4223-x. Epub 2016 Jun 28. PMID 27351548
- [Background] Larsson R, Bernhardsson S, Nordeman L. Effects of eccentric exercise in patients with subacromial impingement syndrome: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2019 Oct 14;20(1):446. doi: 10.1186/s12891-019-2796-5. PMID 31610787
- [Background] O'Sullivan K, McAuliffe S, Deburca N. The effects of eccentric training on lower limb flexibility: a systematic review. Br J Sports Med. 2012 Sep;46(12):838-45. doi: 10.1136/bjsports-2011-090835. Epub 2012 Apr 20. PMID 22522590
- [Background] Talbott And NR, Witt DW. In vivo measurements of humeral movement during posterior glenohumeral mobilizations. J Man Manip Ther. 2016 Dec;24(5):269-276. doi: 10.1179/2042618615Y.0000000007. PMID 27956820
- [Background] Celik D. Comparison of the outcomes of two different exercise programs on frozen shoulder. Acta Orthop Traumatol Turc. 2010;44(4):285-92. doi: 10.3944/AOTT.2010.2367. PMID 21252605
- [Background] Current management of shoulder adhesive capsulitis: a randomized, triple-blind placebo-controlled trial Riyadh a. Almashni1*, abdullah w. Calacattawi2, meshal a. Almeshal3, elaf j. Alsharif4, mohamad w. Hijazi5, shahd a. Abdulwahab5, anfal j. Alsharif6, nasser o. Altufayl7, anwar a. Alghamdi1, hisham a. Almuzayyen
- [Background] Ekelund AL, Rydell N. Combination treatment for adhesive capsulitis of the shoulder. Clin Orthop Relat Res. 1992 Sep;(282):105-9. PMID 1516300
- [Background] Aldon-Villegas R, Ridao-Fernandez C, Torres-Enamorado D, Chamorro-Moriana G. How to Assess Shoulder Functionality: A Systematic Review of Existing Validated Outcome Measures. Diagnostics (Basel). 2021 May 8;11(5):845. doi: 10.3390/diagnostics11050845. PMID 34066777
- [Result] Hollmann L, Halaki M, Kamper SJ, Haber M, Ginn KA. Does muscle guarding play a role in range of motion loss in patients with frozen shoulder? Musculoskelet Sci Pract. 2018 Oct;37:64-68. doi: 10.1016/j.msksp.2018.07.001. Epub 2018 Jul 6. PMID 29986193
- [Result] Raven EE, Haverkamp D, Sierevelt IN, van Montfoort DO, Poll RG, Blankevoort L, Tak PP. Construct validity and reliability of the disability of arm, shoulder and hand questionnaire for upper extremity complaints in rheumatoid arthritis. J Rheumatol. 2008 Dec;35(12):2334-8. doi: 10.3899/jrheum.080067. Epub 2008 Nov 1. PMID 19004045
- [Result] Wee CC, Davis RB, Hamel MB. Comparing the SF-12 and SF-36 health status questionnaires in patients with and without obesity. Health Qual Life Outcomes. 2008 Jan 30;6:11. doi: 10.1186/1477-7525-6-11. PMID 18234099
- [Result] Millar AL, Lasheway PA, Eaton W, Christensen F. A retrospective, descriptive study of shoulder outcomes in outpatient physical therapy. J Orthop Sports Phys Ther. 2006 Jun;36(6):403-14. doi: 10.2519/jospt.2006.2101. PMID 16776489
- [Result] Werner BC, Holzgrefe RE, Griffin JW, Lyons ML, Cosgrove CT, Hart JM, Brockmeier SF. Validation of an innovative method of shoulder range-of-motion measurement using a smartphone clinometer application. J Shoulder Elbow Surg. 2014 Nov;23(11):e275-82. doi: 10.1016/j.jse.2014.02.030. Epub 2014 Jun 9. PMID 24925699
- [Result] Use of smart phone for measuring shoulder rotational range of motion in patients with frozen shoulder: A comparative study Kartik Shah, Mangala Deshpande Priyesha Ramteke Jyoti Singh Anjali Sondawle

DOCUMENTS (1):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT05466435/Prot_000.pdf